CLINICAL TRIAL: NCT06921590
Title: A Randomized, Balanced, Phase 1, Multiple-dose, Open-label, Two-treatment, Two-period, Two-sequence, Crossover, Relative Bioavailability Study to Investigate Lithium Brain/Plasma Pharmacokinetics and Safety of an AL001 Oral Capsule Compared to a Marketed Immediate-release Lithium Carbonate Capsule in Healthy Adult Subjects
Brief Title: A Study to Investigate Lithium Brain/Plasma Pharmacokinetics and Safety of an AL001 Oral Capsule Compared to a Marketed Immediate-release Lithium Carbonate Capsule in Healthy Adult Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alzamend Neuro, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AL001-ALZ03
Record Dates: First submitted 2025-03-19; First posted 2025-04-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-04

CONDITIONS: Pharmacokinetics; Neurology
Keywords: Healthy Controls
MeSH Terms: interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: AL001 then Lithium Carbonate (Other): Participants take 1050 mg of AL001 TID for 14 days then after a washout period, take 150 mg TID of Lithium Carbonate for 14 days.
  Interventions: Drug: AL001; Drug: Lithium Carbonate Capsule
- Sequence 2: Lithium Carbonate then AL001 (Other): Participants take 150 mg of Lithium Carbonate TID for 14 days, then after a washout period, take 1050 mg of AL001 TID for 14 days.
  Interventions: Drug: AL001; Drug: Lithium Carbonate Capsule

INTERVENTIONS:
Drug: AL001 — Crystalized Lithium
  Other Names: lithium salicylate/L-proline cocrystal
Drug: Lithium Carbonate Capsule — Lithium Carbonate

SUMMARY:
The goal of this clinical trial is to assess the safety and effects of a crystalized form of lithium, AL001, when compared to commonly used Lithium Carbonate in healthy volunteers. The main questions this study aims to answer are:

How safe and effective is AL001 when compared to Lithium Carbonate? How is AL001 broken down in the brain and body compared to Lithium Carbonate?

Participants will be asked to:

* Take both the study drug (AL001) and Lithium Carbonate each for a period of 14 days
* Stay overnight at MGH's research unit for two separate 2-week periods
* Participate in two separate 24 hour periods of multiple MRIs and blood draws

DETAILED DESCRIPTION:
This study is researching the effects of a new type of crystalized lithium, AL001, on it's ability to reach the brain and have an effect. The investigators will be comparing this to a commonly used type of lithium, lithium carbonate. Investigators want to see if the crystalized lithium can have the same or better effect when compared to lithium carbonate. Past research has shown a greater effect within the body with crystalized lithium when compared to commonly used lithium.

This past research suggests that crystallized lithium may be more effective, potentially allowing for lower doses and fewer side effects. If successful, this new form of lithium could offer a new and safe treatment option for psychiatric and neurological disorders.

This study involves two, 2-week long overnight stays at the main campus of Massachusetts General Hospital. During these stays participants will receive lithium carbonate for one stay and the crystalized lithium for the other. There are frequent blood draws and brain MRI scans during two periods of the study to look at how the crystalized lithium is broken down in the body and to see how it reaches the brain. This study will compare AL001 to a study reference treatment of lithium carbonate. The majority of the blood draws and MRIs will occur over a 24 hour period during each 2-week long overnight stay at MGH.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects ≥18 and <65 years old in reasonably good physical and psychological health as determined by the Investigator's review of medical and surgical history, physical examination (including neurological examination), 12-lead ECG, vital signs, and clinical laboratory tests.
2. Assessment of subject's mental health status will be conducted to avoid enrolling subjects who are on the verge of a manic or depressive episode. Affective stability, defined by a Young Mania Rating Scale (YMRS) rating of <8 and a Hamilton Depression Rating Scale (HRSD-17) rating of ≤7 at screening and baseline. Assessment of subject's suicidal ideation and behavior (SI/B) using the Columbia-Suicide Severity Rating Scale (C SSRS) will be conducted to avoid enrolling subjects with concerning results, defined as a lifetime history of a suicide attempt, past year level 4 or higher suicidal ideation on the C-SSRS, or past month suicidal ideation of any kind. The "Lifetime/Recent" version will be used at screening and the "Since Last Visit" version will be used subsequently.
3. Able to understand and follow instructions during the study as determined by the Investigator.
4. Willing to follow study procedures.
5. Willing and able to adhere to study restrictions and to be confined at the clinical research center per protocol requirements.
6. Any gender, race, or ethnicity.
7. Able to understand and provide written informed consent.
8. Males (non-vasectomized and vasectomized) must agree to use barrier contraception during the study until after Treatment Period 2 in-clinic follow-up visit on Day 23 (P2).
9. Females must meet one the of the following criteria:

   Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:
   1. Abstinence from heterosexual intercourse from the Screening visit through to at least 30 days after the last dose of the second study drug on Day 14 (P2).
   2. One of the following highly-effective contraceptive methods, used from at least 28 days prior to the Screening visit through to at least 30 days after the last dose of the second study drug on Day 14 (P2).

   i. Systemic contraceptives (combined birth control pills, injectable/implant/ insertable hormonal birth control products, or transdermal patch).

   ii. Intrauterine device (with or without hormones). iii. Male partner vasectomized at least 6 months prior to the Screening visit. c. One of the following double-barrier contraceptive methods, used from the Screening visit through to at least 30 days after the last dose of the second study drug on Day 14 (P2): i. Male condom used simultaneously with diaphragm plus spermicide. ii. Male condom used simultaneously with cervical cap plus spermicide. Or Is of non-childbearing potential, defined as surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation), or is in a postmenopausal state (i.e., at least 1 year without menses prior to the Screening visit).
10. Able to communicate in English, including speaking, reading, and writing.
11. Body mass index (BMI) within 18.0 to 30.0 kg/m2, inclusive, and body weight of at least 50 kg at the time of Screening.
12. ECG recording, after at least 5 minutes of rest in a supine position without clinically significant abnormalities as determined by the Investigator.

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical examination, vital sign measurements, ECG findings, or clinical laboratory findings (as determined by the Investigator) that may affect the safety or successful participation of the subject. Specifically, evidence of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, dermatologic, muscular, or allergic disease or disorder (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) that may affect the safety or successful participation of the subject. Any history of drug hypersensitivity, asthma (with the exception of childhood asthma), urticaria or other severe allergic diathesis.
2. Presence or history of any disorder that may prevent the successful completion of the study.
3. Other severe acute, chronic, or historical medical or psychiatric condition or laboratory abnormality or social circumstance that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
4. History of seizure disorder and/or severe head trauma (other than a single childhood febrile seizure).
5. History or presence of gastrointestinal disease including chronic gastritis, peptic ulcers, inflammatory bowel disease, hemorrhagic gastritis, or duodenitis.
6. History or presence of acute or chronic liver disease as determined by the Investigator.
7. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the study treatments.
8. Any history of frequent headache or migraine.
9. Kidney disease (eGFR <60 mL/minute/1.73 m2).
10. Uncontrolled tachy/brady arrhythmias, atrial fibrillation, or coronary heart failure.
11. Systemic related exclusions:

    1. Active cancer (except squamous cell and basal skin cancers) requiring chemo- or radiation therapy.
    2. Positive test results for HIV, HBV, or HCV (unless quantitative PCR negative for HCV) at Screening.
    3. Uncontrolled hypertension with a sustained blood pressure >160/100 mmHg at Screening, or at check-in on Day -1 (P1).
    4. Fever (body temperature >101.4°F [38.5°C]), acute upper respiratory, or any other infections at Screening, or at check-in on Day -1 (P1).
12. Psychiatric or neurological illnesses (e.g., depression, schizophrenia or other psychotic syndromes, Parkinson's disease and related movement disorders, seizure disorder, and myasthenia gravis).
13. Treatment with haloperidol, antipsychotics, monoamine oxidase inhibitors, neuromuscular blocking agents. Subjects who have ever received immunosuppressant treatment (excluding topical or oral corticosteroids taken 1 and 5 years before Screening, respectively).
14. Hyponatremia, defined as serum sodium laboratory value outside the standard reference range.
15. The use of any medication on a chronic basis with the exception of hormonal contraceptives for females of childbearing potential. An appropriate drug free period will be required for prescription or over the counter (OTC) drugs to washout, particularly of any especially long half-life drugs (see exclusion criteria 16 and 17 below for relevant details).
16. Use of any medication (OTC, prescription medication, vitamins, and herbal supplements) within 14 days prior to the Screening visit and 14 days prior to Day -1 (P1) - or at least 6 times the respective elimination half-life rather than 14 days, whichever is longer - through the completion of the second study drug treatment on Day 14 (P2). Contraception may be continued. Acetaminophen may be concomitantly used at the discretion of the Investigator (up to 1000 mg per day). Non-medicated opthalmic products (for lubrication and comfort) may also be permitted at the discretion of the Investigator. (Section 5.7.10).
17. Prescribed or OTC use of a salicylate-containing product other than low dose aspirin for cardioprotection (e.g., aspirin, magnesium salicylate, bismuth sub-salicylate, salicylazosulfapyridine [sulfasalazine]) from 1 week before first dose of the first study drug on Day 1 (P1) to 1 week after last dosing of the second study drug on Day 14 (P2); any other prescribed anticoagulant medication. (Section 5.7.10).
18. Willingness to refrain from consumption of poppy seeds or quinine (tonic water) 48 hours prior to Day 1 (P1) and throughout the course of the study.
19. Aspirin/nasal polyposis/asthma syndrome.
20. Female who is breastfeeding.
21. Female who is pregnant according to the pregnancy test at Screening or prior to the first dosing of the first study drug on Day 1 (P1); female planning to become pregnant during the study.
22. History of adverse or hypersensitivity reaction to lithium, aspirin, salicylate, L-proline, or any investigational or reference article excipient.
23. Drug/alcohol abuse:

    1. History of drug abuse (barbiturate, amphetamine, benzodiazepine, cocaine, opiates and cannabis) within the last 12 months or a positive urine drug screen at Screening or Day -1 (P1).
    2. Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements or positive ethanol (alcohol) test at Screening or Day -1 (P1).
    3. More than moderate current alcohol consumption. Subjects will be advised to consume no more than 2 units of alcohol per day and completely abstain from 72 hours prior to any visit (1 unit is equal to approximately 10 g of pure alcohol, [250 mL] of beer [5%], 1 small glass [100 mL] of wine [12%], or 35 mL of spirits [35%]).
24. Demonstrating excess xanthine consumption (e.g., ingests more than 5 cups of coffee or equivalent per day). The subject is not willing to refrain from xanthine products for 48 hours prior to check-in on Day -1 (P1). Also, subject is not willing to refrain from grapefruit, pomelo, Seville orange products or juice within 14 days prior to check-in on Day -1 (P1) until discharge from Period 2 treatment on Day 15 (P2).
25. Participation in a clinical trial and receipt of an investigational medication within 30 days or 5 half-lives (if known), whichever is greater, prior to the first dose of the current study drug.
26. History of untreated thyroid dysfunction (due to potential lithium drug-disease interaction).
27. Screening magnetic resonance imaging (MRI)-related exclusion criteria: intracranial mass, evidence of other anatomical findings that might affect safety or causes of cognitive/behavioral impairment as assessed by a qualified neurologist. Subjects must not have any implantable medical device (e.g., aneurysm clip, vagus nerve stimulator, cardiac pacemaker) or be reliant on a removable medical device (e.g., insulin pump) unless that device is certified as MRI compatible. Known intolerability to MRI neuroimaging procedures.
28. Subjects with any past apparent suicide attempt or suicidal behavior, including those with a lifetime history of suicide attempt(s) or a past year level 4 or higher SI/B or past month SI/B (C-SSRS) of any kind.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate differences in brain and/or brain structure lithium PK relative to plasma PK for AL001 capsule compared to a lithium carbonate capsule. | From time zero to the end of the 24 hour 3-dose interval at steady state
  • Brain (and brain structures)-to-plasma ratios between AL001 and lithium carbonate for steady-state PK measures/ parameters
  Area under the plasma and brain concentration versus time curves (AUC) will be measured.
To evaluate differences in brain and/or brain structure lithium PK relative to plasma PK for AL001 capsule compared to a lithium carbonate capsule. | From time zero to the end of the 24 hour 3-dose interval at steady state
  • Similarities and differences between steady state brain and brain structures lithium PK measures/parameters for AL001 and lithium carbonate
  Area under the plasma and brain concentration versus time curves (AUC) will be measured.
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to end of follow-up period at Day 42
  Proportion of participants with adverse events and serious adverse events
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to Day 23 (P2)
  Proportion of participants with abnormal vital signs (from baseline to Day 23 (P2))
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to Day 23 (P2)
  Proportion of participants with abnormal values and change from baseline reading for each ECG parameter. Individual parameters including heart rate, PR, QT, QTcF, QRS, and RR intervals will be collected.
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to Day 23 (P2)
  Proportion of participants with abnormal findings on physical exam.
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to Day 23 (P2)
  Proportion of participants with abnormal values and changes from baseline for each Safety laboratory test (standard hematology, blood chemistry [clinical chemistry], urinalysis, and pregnancy test [for females of childbearing potential only).
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to Day 23 (P2)
  Proportion of participants with prevalence of plasma lithium concentrations above 1.2 mEq/L.
To evaluate the safety and tolerability of AL001 under multiple-dose, steady-state conditions in healthy adult subjects under the conditions of this study. | From enrollment to Day 23 (P2)
  Proportion of participants with prevalence of plasma salicylate concentrations above 30 mg/dL

SECONDARY OUTCOMES:
To characterized AL001 salicylate PK under the conditions of this study | From time zero to the end of the 24 hour 3-dose interval at steady state.
  • Brain (and brain structures)-to-plasma ratios between AL001 and lithium carbonate for steady-state PK measures/ parameters
  Area under the plasma and brain concentration versus time curves (AUC) will be measured.
To characterized AL001 salicylate PK under the conditions of this study | From time zero to the end of the 24 hour 3-dose interval at steady state.
  • Similarities and differences between steady state brain and brain structures lithium PK measures/parameters for AL001 and lithium carbonate
  Area under the plasma and brain concentration versus time curves (AUC) will be measured.
Exploring Brain Pharmacodynamics using Magnetic Resonance Spectroscopy | From Screening (Day 1) to Day 23 (P2)
  Magnetic resonance spectroscopy (MRS) techniques will be applied to explore brain metabolism, including possible metabolic similarities/differences between treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT06921590/ICF_001.pdf